CLINICAL TRIAL: NCT01872091
Title: Analysis of Neuromuscular, Circulatory and Biomechanical Responses After Cryotherapy by Immersion of the Forearm
Brief Title: Analysis of Neuromuscular, Circulatory and Biomechanical Responses After Cryotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: U1111-1143-3579
Record Dates: First submitted 2013-05-27; First posted 2013-06-07 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Healthy Individuals
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cryotherapy by immersion (Experimental): Cryotherapy group immersion (GI) composed of 20 volunteers, which will be subjected to immersion cryotherapy upper limb dominant in cold water (6°C ± 2°C), at the level of the elbow joint.
  Interventions: Other: cryotherapy by immersion
- Control group (Experimental): (CG) consisted of 20 volunteers, which will be submitted to immersion of the dominant upper limb in water at room temperature indifferent to the level of the elbow joint;
  Interventions: Other: Control group

INTERVENTIONS:
Other: cryotherapy by immersion
  Arms: cryotherapy by immersion
Other: Control group
  Arms: Control group

SUMMARY:
Cryotherapy is a resource applied thermal rehabilitation in order to reduce skin temperature and muscle as well as nerve conduction velocity, and promotes vasoconstriction of arteries and veins resulting in decreased blood flow.

DETAILED DESCRIPTION:
Cryotherapy is a resource applied thermal rehabilitation in order to reduce skin temperature and muscle as well as nerve conduction velocity, and promotes vasoconstriction of arteries and veins resulting in decreased blood flow. Thus, this study aims to evaluate neuromuscular and biomechanical assess hemodynamic and autonomic cardiovascular, and investigate the occurrence of changes in conduction velocity due to the superficial blood cryotherapy by immersion of the forearm. The study will be conducted in 40 volunteers, female, between 18 and 30 years, university, healthy. They will be divided into two groups of 20 volunteers, the group immersion cryotherapy (GI) and control group (CG). For immersion cryotherapy group (GI), individuals will be the right arm to the elbow immersed in a container of water at 6°C ± 2°C for 15 minutes. In the control group (CG), volunteers will remain at rest with the right arm in the same position within a vessel containing water at a temperature indifferent for the same period of 15 minutes. The temperature analysis is performed using a infrared thermographer, muscular strength and synergism will be evaluated by a load cell connected to the electromyograph to examine muscle activation of wrist flexors and extensors, serratus anterior, upper and middle trapezius. The records beat to beat blood pressure and heart rate for cardiovascular autonomic and hemodynamic evaluation will be carried out by means of equipment and Finometer electrocardiogram, respectively, before and after application of cryotherapy. In turn, the data of blood flow velocity will be collected by means of Doppler Ultrasound. The results will be processed and analyzed using descriptive statistics, submitted to a linear regression model with mixed effects (fixed and random effects), with p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals, age range: 18 - 30 years old

Exclusion Criteria:

* not present: previous circulatory, nervous or metabolic diseases, metal implants in areas to be studied; fracture on upper limb studied; history of pain or injury in the joints studied
* are not in menstrual period or a week before it
* not be making use of antipyretic drugs

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the strength and muscle synergism after cryotherapy immersion | 2 years
  The objective of this study is to Evaluate the strength and muscle synergism between wrist flexors and extensors after forearm immersion cryotherapy. Testing grip strength will be carried out 3 times in a row, with 4 seconds of maximum voluntary isometric contraction, with a 1 minute interval between them; before, immediately after, 25 minutes and 50 minutes after immersion. Strength evaluation is conducted using a load cell. Concurrent with this test, the signal will be collected electromyographic extensor and flexor wrist, upper and middle trapezius fibers and anterior serratus.

SECONDARY OUTCOMES:
Blood flow velocity before and after immersion of the forearm cryotherapy | 2 years
  The data of blood flow velocity will be collected through the portable Doppler ultrasound wave continues. Immediately before the strength tests will be collected the data from the radial artery blood flow (3 times per collection), so there are no changes due to muscular work required in the handgrip test.

OTHER OUTCOMES:
Changes in skin temperature before and after cryotherapy by immersion of the forearm | 2 years
  The skin temperature data will be acquired by a digital infrared thermographer. Immediately before the strength tests will be collected temperature data cutaneous (3 times per collection), so there are no changes due to muscular work required in testing grip.

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Guirro, Professor, Study Director — University of Sao Paulo
Locations (1):
- Rinaldo Roberto de Jesus Guirro, Ribeirão Preto, São Paulo, Brazil